CLINICAL TRIAL: NCT01077882
Title: Analysis of the Quality of Life, the Clinical Effectiveness and Cost-effectiveness of a Novel Educational Programme in Patients With Psoriasis and Atopic Dermatitis
Acronym: OnderHUIDs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009/691
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: Moderate and severe psoriasis and atopic dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- current therapy (Placebo Comparator)
  Interventions: Other: no educational program
- current therapy with educational program (Experimental)
  Interventions: Behavioral: education on skin disease conditions; Behavioral: Stress-reduction techniques; Behavioral: Lifestyle factors and psycho-education

INTERVENTIONS:
Behavioral: education on skin disease conditions — information about several skin diseases skin function recommendation on care of skin
  Arms: current therapy with educational program
Behavioral: Stress-reduction techniques — Physical Training yoga mindfulness-based stress reduction
  Arms: current therapy with educational program
Behavioral: Lifestyle factors and psycho-education — by dietician and psychiatrist
  Arms: current therapy with educational program
Other: no educational program — standard care without educational program
  Arms: current therapy

SUMMARY:
'OnderHUIDs' is an educational program (Department of Dermatology, University Hospital, Gent) for patients with psoriasis and atopic dermatitis. We want to stimulate the patient to actively participate in their therapeutic approach by enhanced self care. We call the hypothesis that this program will help the patients learn to cope with their disease and to be loyal to their treatment, which will result in a better quality of life, better clinical outcome and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Women or men of any race
* Patients who are 18-75 years of age
* Diagnosis of psoriasis or atopic dermatitis

Exclusion Criteria:

* Patients with a cognitive disorder (not able to understand, speak, read or write..)
* Patients with a significant underlying medical cause (i.e. severe infection, haematologic disease, malignity, severe renal or hepatic disease, major depression) in the last 3 months
* Patients under experimental pharmaceutical medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of a novel educational program on the quality of life and the clinical outcome. | At 12 weeks, after 6 and 9 months
  Therefore quality of life questionnaires are completed at the beginning of the program, at the end of the program (12 weeks), after 6 months and after 9 months. The quality of life questionnaires are Daily life quality index, Skindex 29, EuroQol -5D, Short Form - 36 , Psoriasis disability index, Quality of Life Index for Atopic Dermatitis.
  The clinical effectiveness is determined by measuring psoriasis area and severity index (PASI) or scoring atopic dermatitis (SCORAD) at the beginning of the program, at the end of the program (12 weeks), after 6 months and after 9 months.

SECONDARY OUTCOMES:
Depression severity | At 12 weeks, 6 months and 9 months
  Beck Depression Inventory (BDI) is a self-completed questionnaire with 21 questions. It is one of the most widely used instruments for measuring depression severity. BDI scores are collected during the four study visits.
Lifestyle | At 12 weeks, 6 months and 9 months
  Patients are queried for changes in smoking behaviour and physical activity monthly. Also, stress is examined during the four study visits,therefore we use the Everyday Problem Checklist.
Medical consumption and cost-effectiveness evaluation | At 12 weeks, 6 months and 9 months
  Medical therapy of patients is divided into: topical therapy, systemic therapy, combination of topical and systemic therapy or no therapy. Patients are asked for changes in medical therapy monthly. Also, medical consumption is followed: costs for medication and doctor visits related to the management of the skin disease. EuroQol-5D (EQ-5D) questionnaires are used as standardised instrument to measure health outcomes. For cost-utility analysis, gain in quality-adjusted life years utilities is plotted against time, using the area under the curve approach (cost in EUR/EQ-5D gain).

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be